CLINICAL TRIAL: NCT04052932
Title: A Phase3, Multicentre, Randomized, Double-Blind, Allopurinol and Placebo-Controlled Study to Evaluate the Efficacy and Safety of SHR4640 Monotherapy in Subjects With Gout
Brief Title: A Study of Evaluating the Efficacy and Safety of SHR4640 in Subjects With Gout
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR4640-301
Record Dates: First submitted 2019-08-06; First posted 2019-08-12 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo once a day, orally, for 12 weeks, followed by SHR4640 treatment to 36 weeks
  Interventions: Drug: Placebo oral tablet
- SHR4640 dose1 (Experimental): SHR4640 dose1 once a day, orally, for 36 weeks
  Interventions: Drug: SHR4640 dose1
- SHR4640 dose2 (Experimental): SHR4640 dose2 once a day, orally, for 36 weeks
  Interventions: Drug: SHR4640 dose2
- Allopurinol (Active Comparator): Allopurinol 300mg (milligram) once a day, Orally, for 36 week
  Interventions: Drug: Allopurinol 300 MG

INTERVENTIONS:
Drug: SHR4640 dose1 — tablets，dose1，QD
  Arms: SHR4640 dose1
Drug: SHR4640 dose2 — tablets，dose2，QD
  Arms: SHR4640 dose2
Drug: Placebo oral tablet — tablets，QD
  Arms: Placebo
Drug: Allopurinol 300 MG — tablets，300mg，QD
  Arms: Allopurinol

SUMMARY:
This study will assess the serum uric acid lowering effects and safety of SHR4640 compared to placebo and Allopurinol in patients with gout

ELIGIBILITY:
Inclusion Criteria:

1. Subject who met 1977 or 2015 ACR (American College of Rheumatology) classification of Gout and has a serum acid ≥ 480 μmol/L at screening;
2. 18 kg/m2 ≤Body mass index (BMI)≤ 35 kg/m2

Exclusion Criteria:

1. Subject who is pregnant or breastfeeding;
2. Alanine aminotransferase or Aspartate aminotransferase or total bilirubin>1.5 upper normal limit;
3. Subject with a positive test for HLA-B*5801;
4. Estimated glomerular filtration rate (MDRD formula) <60ml/min;
5. HbA1c>8%;
6. Subject with known hypersensitivity or allergy to SHR4640 and allopurinal, or any component of SHR4640;
7. Subject with kidney stones or suspicion of kidney stones;
8. Subject who has acute gout flares within 2 weeks before randomization;
9. Subject with a history of malignancy within the previous 5 years;
10. Subject with a history of active peptic ulcer within a year;
11. Subject with a history of xanthine urine.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 594 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with a serum uric level≤360μmol/l. | Week 12
  Proportion of subjects with a serum uric level≤360μmol/l.

SECONDARY OUTCOMES:
Proportion of subjects with a serum uric level≤360μmol/l | Week 36
  Proportion of subjects with a serum uric level≤360μmol/l
Percentage change from baseline in serum uric level | Up to 36 weeks
  Percentage change from baseline in serum uric level
Actual change from baseline in serum uric level | Up to 36 weeks
  Actual change from baseline in serum uric level
Proportion of subjects with a serum uric level≤360μmol/l | Up to 36 weeks
  Proportion of subjects with a serum uric level≤360μmol/l

CONTACTS AND LOCATIONS:
Overall Officials: Chunde Bao, Principal Investigator — RenJi Hospital
Locations (1):
- RenJi Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided